CLINICAL TRIAL: NCT01752725
Title: Comparison of BiCision® Versus UltraCision® During Laparoscopic Supracervical Hysterectomy (LASH): A Prospective, Controlled, Randomized, Non-inferiority in Vivo Human Study.
Brief Title: Comparison of BiCision® Versus UltraCision® During Laparoscopic Supracervical Hysterectomy (LASH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Erbe Elektromedizin GmbH (Industry)
Responsible Party: Principal Investigator, Bernhard Kraemer, Executive / Investigator, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04122012
Record Dates: First submitted 2012-12-04; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Uterine Bleeding Disorders; Benign Uterine Conditions; Focus: Comparison of Two Instruments
Keywords: supracervical hysterectomy; vessel sealing; bipolar electrocoagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BiCision Arm (Experimental): Coagulation with BiCision
  Interventions: Device: BiCision®
- Ultracision Arm (Active Comparator): Coagulation with Ultracision
  Interventions: Device: Ultracision® Har-monic Scalpel(Ethicon)

INTERVENTIONS:
Device: BiCision®
  Arms: BiCision Arm
Device: Ultracision® Har-monic Scalpel(Ethicon)
  Arms: Ultracision Arm

SUMMARY:
The aim of the study is the evaluation of the efficiency and safety of the new, CE-certified thermofu-sion and dissection instrument BiCision® in comparison with the long established Ultracision® Har-monic Scalpel(Ethicon)during a laparoscopic supracervical hysterectomy (LASH).

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* gender: female
* indication for laparoscopic supracervical hysterectomy with no adnexectomyor other surgery
* will and the capability to comply the study requirements
* signed informed consent

Exclusion Criteria:

* Invasive malignome in the pelvis
* Cardiac pacemaker or implanted defibrilator if no informations are available about the compatibil-ity with RF energy
* Abnormal blood parameters (values less than factor 0.8 or more than 1.25 compared to the val-ues of creatinine and standard hemogram)
* Abnormal coagulation parameters: PTT > 40 sec. and / or Quick's-Value< 50% (the use of antiplateletsup to a max. of 100mg/d is no exclusion criteria)
* Inability to understand the purpose of the study
* status after a laparotomy by a longitudinal incision
* intraabdominal adhesions (at the beginning of the surgery ≥ 5 sectioning for adhesiolysis)
* open laparoscopy required
* different anatomical situations that yields to different surgery requirements
* conspicuous PAP, cervixmyoma or endometriosis of the rectovaginale space

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Operation time | Participants will be followed for the duration of hospital stay, an expexted average of 8 months
  The primary objective is the operation time for each preparation side and instrument needed from the beginning of the removal of the cornual structure of the uterus (uterine cornu) till the completely removal of the parametric tissue directly before removal of the corpus uteri from the cervix.

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Wallwiener, Professor, Study Chair — University Hospital Tuebingen; Bernhard Krämer, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital, Tübingen, Germany